CLINICAL TRIAL: NCT00419406
Title: Medium-Dose UVA1 Versus Narrow-Band UVB Phototherapy: A Randomized Double-Blind Controlled Cross-Over-Study
Brief Title: Medium-Dose UVA1 Versus Narrow-Band UVB in Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Dr. Thilo Gambichler, Department of Dermatology, Ruhr University of Bochum
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2466
Record Dates: First submitted 2007-01-04; First posted 2007-01-08 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Atopic Dermatitis
Keywords: UVA1; N-B UVB; phototherapy; atopic dermatitis; SCORAD index
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: UVA1 (Experimental)
  Interventions: Procedure: UVA1 phototherapy
- B: NB UVB (Experimental)
  Interventions: Procedure: NB-UVB phototherapy

INTERVENTIONS:
Procedure: UVA1 phototherapy
  Arms: A: UVA1
Procedure: NB-UVB phototherapy
  Arms: B: NB UVB

SUMMARY:
Atopic dermatitis (AD) is a very common disorder that is characterized by pruritic inflammatory skin lesions, with patients usually having an individual or family history of atopic diseases in their background. Phototherapy is among the first-line approaches in the management of AD. In this context, a variety of studies have shown a beneficial effect of natural or artificial UV radiation in atopic dermatitis (AD). The past ten years have seen the introduction of new phototherapeutic regimens for AD, including UVA1 and NB-UVB.UVA1 seems to be more effective than the above mentioned broadband spectra, in particular in acute severe AD. The aim of the present study is the comparison of UVA1 and NB-UVB phototherapy in the treatment of AD. Additionally, the course of several cytokines, human beta-defensins, and SMAD-proteins will be evaluated during the course of treatment.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a very common disorder that is characterized by pruritic inflammatory skin lesions, with patients usually having an individual or family history of atopic diseases in their background (e.g., allergic asthma and rhinitis). Defective skin barrier, immunological dysfunctions (type I and IV allergy), genetic disorders, and psychological factors contribute to the pathogenesis of AD. However, among these factors, CD4+ Th cells are reported to play a particularly crucial role in the pathogenesis of AD. Phototherapy is among the first-line approaches in the management of AD. In this context, a variety of studies have shown a beneficial effect of natural or artificial UV radiation in atopic dermatitis (AD). Different broadband UV spectra (BB-UVA, BB-UVB, BB-UVA/BB-UVB) and combined treatment modalities such as balneophototherapy and PUVA have previously been proven to be effective in AD. However the past ten years have seen the introduction of new phototherapeutic regimens for AD, including UVA1 and NB-UVB.UVA1 seems to be more effective than the above mentioned broadband spectra, in particular in acute severe AD. The aim of the present study is the comparison of UVA1 and NB-UVB phototherapy in the treatment of AD. Additionally, the course of several cytokines, human beta-defensins, and SMAD-proteins will be evaluated during the course of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic AD (Hanifin and Rajka, 1980); moderate to severe disease with SCORAD-index > 30 (maximum = 102).
* Age > 18 years
* No topical steroids (except 1% hydrocortisone) or topical/systemic antibiotics or antihistamines within the last 2 weeks, no systemic glucocorticosteroids or other immunosuppressive agents within the last 8 weeks, no phototherapy within the last 12 weeks before inclusion

Exclusion Criteria:

* Pregnancy or lactation
* Skin cancer or dysplastic naevi, photosensitive skin diseases, autoimmune diseases or relevant cardiovascular diseases
* Photo-skin type I according to Fitzpatrick

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Clinical improvement during UVA1/NB-UVB phototherapy using a validated
SCORAD index

SECONDARY OUTCOMES:
Comparison of efficacy between UVA1 and NB-UVB phototherapy using a validated
SCORAD index

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Gambichler, MD, Principal Investigator — Department of Dermatology, Ruhr University Bochum; Alexander Kreuter, MD, Principal Investigator — Department of Dermatology, Ruhr University Bochum
Locations (1):
- Department of Dermatology, Ruhr University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Gambichler T, Tomi NS, Skrygan M, Altmeyer P, Kreuter A. Alterations of TGF-beta/Smad mRNA expression in atopic dermatitis following narrow-band ultraviolet B phototherapy: results of a pilot study. J Dermatol Sci. 2006 Oct;44(1):56-8. doi: 10.1016/j.jdermsci.2006.06.004. Epub 2006 Aug 4. No abstract available. PMID 16889943
- [Result] Gambichler T, Skrygan M, Tomi NS, Altmeyer P, Kreuter A. Changes of antimicrobial peptide mRNA expression in atopic eczema following phototherapy. Br J Dermatol. 2006 Dec;155(6):1275-8. doi: 10.1111/j.1365-2133.2006.07481.x. PMID 17107401
- [Result] Gambichler T, Othlinghaus N, Tomi NS, Holland-Letz T, Boms S, Skrygan M, Altmeyer P, Kreuter A. Medium-dose ultraviolet (UV) A1 vs. narrowband UVB phototherapy in atopic eczema: a randomized crossover study. Br J Dermatol. 2009 Mar;160(3):652-8. doi: 10.1111/j.1365-2133.2008.08984.x. Epub 2008 Dec 11. PMID 19120333